CLINICAL TRIAL: NCT05534568
Title: A Randomized Controlled Trial of the Parent-Child Assistance Program in Oklahoma
Brief Title: The Oklahoma Parent-Child Assistance Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: University of Oklahoma Outreach (Unknown); Oklahoma Mental Health and Substance Abuse (Unknown); Arnall Family Foundation (Unknown); Oklahoma Human Services (Unknown); OU Dodge Family College of Arts and Sciences (Unknown); Casey Family Programs (Unknown); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14394
Record Dates: First submitted 2022-06-08; First posted 2022-09-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Substance Use Disorders; Pregnancy Related; Alcohol Use Disorder (AUD); Alcohol Use Complicating Pregnancy, First Trimester; Alcohol Use Complicating Pregnancy, Second Trimester; Alcohol Use Complicating Pregnancy, Third Trimester; Alcohol Use Complicating Pregnancy, Unspecified Trimester; Alcohol Use Complicating Pregnancy, Childbirth, and the Puerperium; Fetal Alcohol Spectrum Disorders; Fetal Alcohol Syndrome; Drug Use Disorders; Drug Use Complicating Pregnancy, First Trimester; Drug Use Complicating Pregnancy, Second Trimester; Drug Use Complicating Pregnancy, Third Trimester; Drug Use Complicating Pregnancy, Unspecified Trimester; Drug Use Complicating Pregnancy, Childbirth, and the Puerperium; Maternal Drugs Affecting Fetus
Keywords: Parent-child assistance; Substance use disorder; addictions; drug dependence; drug abuse; alcohol dependence; alcohol abuse; alcoholism; recovery services; PCAP
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Fetal Alcohol Spectrum Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group consists of women who have used alcohol, opioids, or other drugs during pregnancy and their children. Mothers who are randomly assigned to the treatment group will receive PCAP services through the work of highly trained, closely supervised case managers.
  Interventions: Other: Parent-Child Assistance Program
- Control Group (No Intervention): The control group consists of women who have used alcohol, opioids, or other drugs during pregnancy and their children. Women in the control group will be provided with a service resource list and receive services as usual, but they will not be enrolled in PCAP.

INTERVENTIONS:
Other: Parent-Child Assistance Program — Case managers work closely with mothers over the course of three years, meeting the mothers in their own homes when possible, to help them to set goals and take advantage of available resources.
  Arms: Treatment Group

SUMMARY:
The Parent-Child Assistance Program (PCAP) helps mothers who have used alcohol, opioids, or other drugs during pregnancy and their children through the work of highly trained, closely supervised case managers. Case managers work closely with mothers over the course of three years, meeting the mothers in their own homes when possible, to help them to set goals and take advantage of available resources. The primary aims of PCAP include: (1) assisting mothers in obtaining substance use disorder (SUD) treatment and staying in recovery, (2) linking mothers to community resources that will help them build and maintain healthy, independent family lives for themselves and their children, and (3) preventing future drug and alcohol use during pregnancy.

This study brings PCAP to Oklahoma (the state with the highest incarceration rate for women, where most enter the criminal justice system for drug charges) for the first time. This five-year project includes 200 women who will enroll in the study and be randomly assigned to the treatment (100 women) or control group (100 women). The intervention (i.e., PCAP services) will take place over a three-year period at two sites: Oklahoma City, Oklahoma and Tulsa, Oklahoma.

This evaluation will measure participants' substance use, substance use disorder (SUD) treatment outcomes, and a host of other well-being outcomes-including but not limited to subsequent substance-exposed births, use of public assistance, education, use of family planning methods, and employment-to evaluate the effects of PCAP services. Among these, the investigators have identified four key outcomes: (1) the mother is on a reliable method of birth control, (2) abstinence for six months, (3) child custody (i.e., placement of children in foster care and/or with kinship providers), and (4) criminal justice involvement.

DETAILED DESCRIPTION:
The Parent-Child Assistance Program (PCAP) helps mothers who have used alcohol, opioids, or other drugs during pregnancy and their children through the work of highly trained, closely supervised case managers. Case managers work closely with mothers over the course of three years, meeting the mothers in their own homes when possible, to help them to set goals and take advantage of available resources. The primary aims of PCAP include: (1) assisting mothers in obtaining substance use disorder (SUD) treatment and staying in recovery, (2) linking mothers to community resources that will help them build and maintain healthy, independent family lives for themselves and their children, and (3) preventing future drug and alcohol use during pregnancy.

This study brings PCAP to Oklahoma (the state with the highest incarceration rate for women, where most enter the criminal justice system for drug charges) for the first time. In Washington state, where PCAP was first developed and implemented by researchers at the University of Washington in 1991 with federal funding, PCAP has expanded to 15 sites, covering 19 counties and a large majority of the state's population. The population the Washington program serves is highly vulnerable with significant childhood trauma. Eighty-nine percent of the mothers themselves had parents who abused alcohol and drugs. Nearly two-thirds were physically or sexually abused as children. Approximately one quarter had spent time in foster care. Thirty-five percent did not have a high school degree. Among 36% of mothers, Temporary Assistance for Needy Families (TANF) was their main source of income. The investigators anticipate that PCAP participants in Oklahoma will share similar characteristics with those in Washington.

PCAP in Washington conducts evaluations focused on tracking outcomes for all participants. Despite the complex needs and vulnerability of this population and the tenuous situation of substance abuse while pregnant, PCAP outcomes are impressive. Among 1,561 graduates of the 3-year program between 2014-2020, at their exit from the program:

* 90% had completed SUD treatment or were in progress
* 82% were abstinent from alcohol and drugs for 6 months or more during the program and/or regularly using reliable contraception
* 54% had attended or completed classes (GED, college, or work training)
* 70% of the mothers had retained or regained legal custody of their child
* 93% had obtained well child visits and were up to date on child immunizations

Graduates of Washington PCAP were also less likely to use illicit drugs and receive TANF and more likely to be employed, use reliable contraceptives, and reside in permanent or stable housing. Furthermore, the Washington State legislature, prior to expanding the program, requested a cost savings analysis. This analysis, based on robust evaluation results, shows that the program likely realizes multiple sources of cost savings from reduced dependence on child welfare, fewer subsequent alcohol- and drug-exposed children, and reduced dependence on public assistance, among other benefits. The investigators expect similar outcomes for PCAP in Oklahoma.

This five-year project includes 200 women who will enroll in the study and be randomly assigned to the treatment (100 women) or control group (100 women). The intervention (i.e., PCAP services) will take place over a three-year period at two sites: Oklahoma City, Oklahoma and Tulsa, Oklahoma. The control group will be provided with a service resource list and receive services as usual but will not be enrolled in PCAP. The intervention will conclude with sufficient time for a six-month follow-up survey for women who are among the first to enroll in PCAP.

The evaluation of Oklahoma PCAP includes multiple surveys to measure participants' substance use, substance use disorder (SUD) treatment outcomes, and a host of other well-being outcomes, including but not limited to subsequent substance-exposed births, use of public assistance, education, use of family planning methods, and employment. Among these, the investigators have identified four key outcomes: (1) the mother is on a reliable method of birth control, (2) abstinence for six months, (3) child custody (i.e., placement of children in foster care and/or with kinship providers), and (4) criminal justice involvement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Women who have used alcohol, opioids, or other drugs during pregnancy
* Women who are (1) pregnant or have a child under 24 months old who was exposed to substances and are not well connected to community services or (2) have a child with fetal Alcohol Spectrum Disorder and are currently with at-risk alcohol use and in childbearing years
* Resides in Oklahoma City, Oklahoma or Tulsa, Oklahoma

Exclusion Criteria:

* Not meeting eligible criteria above
* Incarcerated at the time of enrollment
* Enrollment in similar services (i.e., ReMerge, Systems of Care (SOC) and/or Family Treatment Courts (FTC) and heading to Termination of Parental Rights (TPR))
* If the participant is receiving services from the Substance use Treatment and Recovery (STAR) Prenatal Clinic and is part of the research, their enrollment in PCAP will be delayed until STAR Prenatal Clinic graduation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in using a reliable method(s) of birth control | Measured every six months up to 4 years
  The mother is on a reliable method(s) of birth control.
Change in abstinence | Measured every six months up to 4 years
  The mother is abstinent from alcohol and drugs for at least six months.

SECONDARY OUTCOMES:
Change in criminal justice involvement | Measured every six months up to 4 years
  The mother has had no new involvement with the criminal justice system.
Change in child custody | Measured every six months up to 4 years
  The mother has physical custody of the index child.
Change in stable housing | Measured every six months up to 4 years
  The mother resides in stable housing.
Change in employment | Measured every six months up to 4 years
  The mother is employed.
Change in education | Measured every six months up to 4 years
  The mother has completed or is enrolled in educational program.
Change in use of public benefits | Measured every six months up to 4 years
  The mother receives public benefits (e.g., housing, food, cash)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Maher, Ph.D., Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - Oklahoma City, Oklahoma City, Oklahoma
  - Tulsa, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher EJ, Stoner SA, Gerlinger J, Ferraro AC, Lepper-Pappan H. Study protocol for a randomized controlled trial of the Parent-Child Assistance Program: a case management and home visiting program for people using substances during pregnancy. Trials. 2024 Apr 16;25(1):264. doi: 10.1186/s13063-024-08098-6. PMID 38627843
- See also: PCAP Website — http://Ou.edu/pcap